CLINICAL TRIAL: NCT05200013
Title: A Phase 1, Multi-Center, Open-Label Study to Assess Safety, Tolerability, Pharmacokinetics, and Preliminary Efficacy of BAT7104 in Patients With Advanced Solid Tumours
Brief Title: BAT7104 in Patients With Advanced Solid Tumours
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bio-Thera Solutions (Industry)
Collaborators: Emerald Clinical Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: BAT-7104-002-CR
Record Dates: First submitted 2021-11-25; First posted 2022-01-20 (Actual); Last update posted 2024-10-18 (Actual); Status verified 2023-10

CONDITIONS: Patients With Advanced Solid Tumors

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Cohort 1 (Experimental): Dose 0.3mg/kg
  Interventions: Biological: BAT7104
- Cohort 2 (Experimental): Dose 1mg/kg
  Interventions: Biological: BAT7104
- Cohort 3 (Experimental): Dose: 3 mg/kg
  Interventions: Biological: BAT7104
- Cohort 4 (Experimental): Dose: 10 mg/kg
  Interventions: Biological: BAT7104
- Cohort 5 (Experimental): Dose: 20 mg/kg
  Interventions: Biological: BAT7104
- Cohort 6 (Experimental): Dose: 40 mg/kg
  Interventions: Biological: BAT7104

INTERVENTIONS:
Biological: BAT7104 — Symmetric IgG-like AntiPD-L1/CD47 Bispecific Antibody Solution for Injection BAT7104 injection available in 100 mg/2 mL (50 mg/mL) dosage

SUMMARY:
This is a prospective multi-centre, Open-Label Study to Assess Safety, Tolerability, Pharmacokinetics, and Preliminary Efficacy of BAT7104 in Patients with Advanced Solid Tumours in Australia.

ELIGIBILITY:
Inclusion Criteria:

1. Able to give voluntary informed consent and understand the study and are willing to follow and complete all the study required procedures.
2. Aged ≥ 18 years
3. Life expectancy ≥ 3 months.
4. Eastern Cooperative Oncology Group （ECOG）performance status ≤ 1.
5. Histologically/cytologically confirmed, locally advanced unresectable or metastatic solid tumours that are refractory to standard therapy, or for whom no standard therapy exists, and where standard therapy is contraindicated or has been declined by the patient. Note that certain malignancies can be included based on imaging (e.g., HCC) and can be included based on the discretion of the PI, Sponsor Medical Monitor approval.
6. Has measurable or evaluable disease per RECIST v1.1. that was not in a prior radiation or other locally treated area, unless imagingbased progression has been clearly documented following radiation or other local therapy.
7. Adequate haematological, liver, and kidney function
8. International normalized ratio (INR) /prothrombin time (PT)< 2, activated partial thromboplastin time (aPTT) ≤ 1.5 × upper limits of normal （ULN）.
9. Must agree to adhere to the current state and national advice regarding minimising exposure to COVID-19 from the first Screening visit until the end of study (90-day follow-up) visit.

Exclusion Criteria:

1. Females who are pregnant or nursing;
2. Receiving concurrent anticancer therapy or investigational therapy (including chemotherapy, radiation therapy, surgery, immunotherapy, hormonal therapy, targeted therapy, biologic therapy);
3. Has remaining AEs > Grade 1 from prior antitumour treatment as per CTCAE v5.0, with the exception of alopecia or ≤ Grade 2 peripheral neuropathy. Patients with chronic Grade 2 toxicities may be eligible per discretion of the Investigator or designee and Sponsor Medical Monitor (e.g., Grade 2 chemotherapy induced neuropathy).
4. Patients with primacy central nervous system (CNS) malignancy, symptomatic CNS metastases, meningeal metastases or leptomeningeal disease are not allowed. Note: Patients with asymptomatic CNS metastases are eligible if clinically controlled, which is defined as 1) ≥4 weeks of stable neurologic function following CNSdirected therapy prior to Cycle 1 Day 1 dosing, 2) no evidence of CNS disease progression as determined by radiographic imaging ≥ 4 weeks prior to Cycle 1 Day 1 dosing, 3) ≥ 2 weeks from discontinuation of anti-seizure and steroid therapies (receiving prednisone ≤ 10mg or equivalent steroid therapies is allowed) prior to Cycle 1 Day 1 dosing.
5. Had major surgery within 28-days of the Screening visit. Note: Patients who have undergone a surgical procedure ≥ 28-days prior to Screening must have recovered adequately from the toxicity and/or complications from the intervention before the first dose of study drugs. Exception: no waiting period applies following port-a-cath placement for venous access.
6. History of tissue or organ transplantation.
7. History of severe infection deemed clinically significant by the PI or designee within 4 weeks or signs and symptoms of any active infection within 2 weeks prior to the first dose of study drugs.
8. History of human immunodeficiency virus (HIV) infection or history of autoimmune diseases.
9. Active hepatitis B or C.
10. History of a Grade 3 or Grade 4 allergic reaction to treatment with another monoclonal antibody.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2022-04-29 (Actual); Primary Completion 2024-06-25 (Actual); Study Completion 2024-06-25 (Actual)

PRIMARY OUTCOMES:
Dose-limiting toxicity (DLT) | A minimum of 28 days after first dose of BAT-7104
  Number of subjects who experience DLT events during 28 days. Toxicity will be graded according to CTCAE, Version 5.0.
Adverse Events (AEs) | up to 90 days after the last dose, an average of 1 year
  Incidence of treatment -related AEs as assessed by CTCAE, Version 5.0.
Serious adverse events (SAEs) | From the time of informed consent to 90 days after the last dose, an average of 1 year
  Any SAE that is judged by the PI or designee to be related to the study medication must be reported regardless of the amount of time since the last dose received. Follow-up information collected for any initial report of an SAE must also be reported to the Sponsor (or its designee) within 24 hours of receipt by the PI or designee.

SECONDARY OUTCOMES:
Cmax (Maximum serum concentration) | up to Cycle 6, each cycle is 14 days
  Maximum observed plasma or serum concentration
Presence of anti-drug antibodies (ADAs) / neutralizing antibodies (NAbs) | up to Cycle 6, each cycle is 14 days
Objective response rate (ORR) | 12 months (anticipated)
  The ORR is defined as the proportion of subjects with confirmed CR or confirmed PR, based on RECIST Version 1.1.
Tmax (Time to reach maximum serum concentration) | up to Cycle 6, each cycle is 14 days
  Time to Maximum concentration
AUC0-inf after Cycle 1 administration and AUC0- λ after Cycle 6 administration | up to Cycle 6, each cycle is 14 days
  area under the serum concentration versus time curve from time zero to infinity and to time λ
Systemic Clearance (CL) | up to Cycle 6, each cycle is 14 days
  Systemic dose clearance
Vss (volume of distribution at steady state) | up to Cycle 6, each cycle is 14 days
  Amount of drug in the body divided by plasma concentration
t1/2 (terminal half-life) | up to Cycle 6, each cycle is 14 days
  Apparent terminal-phase disposition half-life.

CONTACTS AND LOCATIONS:
Locations (2):
- Australia (2):
  - Macquarie University, Sydney, New South Wales
  - One Clinical Research Pty Ltd, Nedlands